CLINICAL TRIAL: NCT05053945
Title: Helicobacter Pylori, Atrophic Gastritis and Intestinal Metaplasia Registry and Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HAR-P Protocol_v1
Record Dates: First submitted 2020-07-14; First posted 2021-09-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Helicobacter Pylori; Atrophic Gastritis; Intestinal Metaplasia
MeSH Terms: conditions — Gastritis, Atrophic | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Esophagogastroduodenoscopy — To set up a prospective study and registry (HAR-P) for patients with H. pylori infection, atrophic gastritis or intestinal metaplasia to evaluate their clinical features and outcomes. The objectives include:
  1. Assess the short- and long-term patient outcomes of H. pylori patients
  2. Characterize factors involved in the progression or regression of pre-neoplastic lesions, namely atrophic gastritis and intestinal metaplasia
  3. Gather information for a better understanding on the efficacy and role of surveillance
  4. Potential for the development of new screening/surveillance strategies and tools for better risk stratification of patients
  5. Establish a biobank for H. pylori, atrophic gastritis and intestinal metaplasia patients

SUMMARY:
Since much is unknown about factors that lead to progression of the pre-neoplastic lesions and cancer. In addition, there is ongoing debate on the optimal surveillance intervals and techniques. To solve these important clinical questions, the establishment of a registry for a longitudinal study is planned.

DETAILED DESCRIPTION:
Helicobacter pylori is believed to affect more than half of the world's population and is thought to affect nearly 2 million people in Hong Kong alone. It is a major cause of peptic ulcer disease and is implicated in the pathogenesis of the majority of gastric cancers. Since 1994, the World Health Organization has designated H. pylori infection as a class 1 carcinogen. Gastric cancer was the sixth commonest malignancy in Hong Kong in 2015; it was also the second commonest cause of death from cancer in Asia. It is thought that chronic inflammation of the gastric mucosa caused by H. pylori progresses to pre-neoplastic lesions, namely atrophic gastritis and intestinal metaplasia, before developing into frank dysplasia and carcinoma. Successful H. pylori eradication can lead to a rapid decrease in active inflammation, with early treatment effective in preventing the progression of disease. It is believed that atrophic gastritis may be reversible, whereas intestinal metaplasia has passed the point of no return and unlikely to have regression. National screening programmes in both Japan and Korea recommend endoscopy for all men and women over 40 years of age with several uncontrolled trials suggesting that this has led to a reduction of mortality due to gastric cancer. However, in countries with a lower incidence of gastric cancer, this population-based approach may not be cost-effective. Much is unknown about factors that lead to progression of the pre-neoplastic lesions and cancer. In addition, there is ongoing debate on the optimal surveillance intervals and techniques. To solve these important clinical questions, the establishment of a registry for a longitudinal study is planned.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years of age
* Written informed consent obtained
* Diagnosed with current or past H. pylori infection,
* Histologically proven atrophic gastritis (body and/or antrum of stomach), intestinal metaplasia (complete and incomplete), dysplasia (any grade) and/or gastric cancer (post- treatment)

Exclusion Criteria:

* Co-morbid illness that prohibit endoscopic surveillance
* Declines for study questionnaire, biobanking of specimens and/or regular review per study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria
  1. Adults >= 18 years of age
  2. Written informed consent obtained
  3. Diagnosed with current or past H. pylori infection,
  4. Histologically proven atrophic gastritis (body and/or antrum of stomach), intestinal metaplasia (complete and incomplete), dysplasia (any grade) and/or gastric cancer (post-treatment)
  Exclusion Criteria
  1. Co-morbid illness that prohibit endoscopic surveillance
  2. Declines for study questionnaire, biobanking of specimens and/or regular review per study protocol
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes of H. pylori patients | 3 years
  Prevalence of H. Pylori, atrophic gastritis, intestinal metaplasia, gastric cancer

SECONDARY OUTCOMES:
Risk factors of gastric pre-cancerous lesions and cancers | 3 years
  Proportion and risk factors for developing gastric pre-cancerous lesions and cancers
Risk factors of atrophic gastirtis | 3 years
  Proportion and risk factors for developing atrophic gastritis
Risk factors of intestinal metaplasia | 3 years
  Proportion and risk factors for developing intestinal metaplasia and progression

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - S.H. Ho Centre for Digestive Health, Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No